CLINICAL TRIAL: NCT03202602
Title: The Benefits of Telemedicine in CPAP Treatment of Obstructive Sleep Apnea Syndrome (OSAS)
Brief Title: Benefits of Telemedicine in CPAP Treatment
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Jenny Theorell-Haglöw, Principal Investigator, Uppsala University
Other Study IDs: TelemedCPAP
Record Dates: First submitted 2017-05-12; First posted 2017-06-28 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Continuous positive airway pressure; Telemoedicine
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telemedicine: Patients randomized to receive telemonitoring in combination with telephone calls after CPAP start.
  Interventions: Other: Telemonitoring of CPAP treatment
- Standard care: Patients randomized to receive usual office visits after CPAP start.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Telemonitoring of CPAP treatment — Telemedicine technology allows for monitoring of CPAP pressure, air leaks, apnea-hypopnea index (AHI) and compliance on a daily basis.
  Groups: Telemedicine
Other: Standard care — Office visits and monitoring of CPAP treatment at each visit.
  Groups: Standard care

SUMMARY:
Continuous positive airway pressure (CPAP) is the first choice of treatment for moderate to severe obstructive sleep apnea syndrome (OSAS). Although adherence is critical for achieving a good treatment effect, and early intervention if treatment problems emerge is important for achieving good adherence, information on patient compliance is usually based on assessment of the first few weeks of treatment. Telemedicine technology allows for monitoring of CPAP pressure, air leaks, apnea-hypopnea index (AHI) and compliance on a daily basis and could therefore be an option allowing for adequate support and quick response if a patient has problems with the treatment. In addition, improving early experiences of CPAP, identifying patients in need of more intensive support could potentially improve adherence but also reduced cost of care, and increased patient satisfaction.

The proposed study will recruit 200 OSAS patients starting CPAP treatment; 100 patients randomized to afterwards receiving telemonitoring in combination with telephone calls, and 100 patients randomized to receiving usual office visits. All patients will in addition answer questionnaires on sleep and health, quality of life, and patient satisfaction after the first CPAP information visit and then again after 6 months of treatment. At time of follow-up all patients will also answer questionnaires on side effects of CPAP. Health economic variables will also be measured throughout the testing period.

The study will provide valuable information regarding benefits of telemonitoring in clinical work with CPAP therapy. Implementation of telemedicine-based monitoring of CPAP therapy may be an important part of increasing adherence among patients but also in the development of a more cost-effective care as it can provide clinics with increased treatment capacity and follow-up of both new and established patients. It would further improve the care for these patients who often have a lifelong treatment, which aims to reduce the risk of developing cardiovascular disease or premature death.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with OSA and scheduled to receive CPAP treatment

Exclusion Criteria:

* Patients not understandning Swedish
* Patients not eligible for CPAP start within a group session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed obstructive sleep apnea syndrome (OSAS) scheduled to receive continuous positive airway pressure (CPAP).
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
CPAP adherence | 6 months
  Time of CPAP use at follow-up. Assesed from count in CPAP machine.

SECONDARY OUTCOMES:
Patient satisfaction regarding CPAP treatment and contact with clinic | 6 months
  Patient satisfaction regarding CPAP treatment and contact with clinic. Assessed via questionnaire.
Number of visits/contacts. | 6 months
  Number of visits/contacts. Assessed via hospital computer records.
Duration of visits/contacts. | 6 months
  Time duration of visits/contacs. Assessed via hospital computer records.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Theorell-Haglöw, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ssegonja R, Ljunggren M, Sampaio F, Tegelmo T, Theorell-Haglow J. Economic evaluation of telemonitoring as a follow-up approach for patients with obstructive sleep apnea syndrome starting treatment with continuous positive airway pressure. J Sleep Res. 2024 May;33(3):e13968. doi: 10.1111/jsr.13968. Epub 2023 Jun 20. PMID 37337981
- [Result] Delijaj F, Lindberg E, Johnsson L, Kristiansson P, Tegelmo T, Theorell-Haglow J. Effects of telemonitoring follow-up, side effects, and other factors on CPAP adherence. J Clin Sleep Med. 2023 Oct 1;19(10):1785-1795. doi: 10.5664/jcsm.10686. PMID 37323036